CLINICAL TRIAL: NCT04726852
Title: Comparison of Arterial Pressure Waveform Derived dp/dt Versus Transesophageal Echocardiogram Derived Left Ventricular dp/dt Max in the Intra-operative Setting
Brief Title: Arterial Pressure vs. TE Echo dp/dt
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 1655978
Record Dates: First submitted 2021-01-21; First posted 2021-01-27 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Myocardial Contraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients having elective cardiac surgery
  Interventions: Device: Concurrent comparison

INTERVENTIONS:
Device: Concurrent comparison — Concurrent comparisons at defined procedure events

SUMMARY:
This study seeks to assess the strength of correlation between arterial pressure waveform derived contractility as quantified by the maximal rate of pressure change ans a function of time (dp/dtmax) and transesophageal echocardiographically (TEE) determined contractility, also quantified by dp/dtmax. In addition, correlations between dp/dtmax. In addition, TEE derived assessment of ejection fraction will provide guidance for relating this new parameter with other standard contractility assessments.

DETAILED DESCRIPTION:
The Hypotension Prediction Index (HPI, Edwards LifeScience, Irvine, CA) software is a new technology that integrates selected dynamic cardiovascular measurements, using the arterial pressure waveform, to predict impending intra-operative hypotensive episodes. In addition, the monitor provides a calculated (dp/dtmax), determined from the radial arterial pressure waveform as a guide to optimal therapeutic interventions. A recent study has demonstrated significant correlation between radial arterial dp/dtmax values calculated with the HPI software to those calculated using echocardiography in patients with acute heart failure in the cardiac ICU setting, especially in those with higher systemic vascular resistance, lower cardiac output, and lower stroke volumes.

This study seeks to assess the strength of these correlations in the intra-operative setting in patients with normal and abnormal cardiac function. Corroboration of the reliability of this newer method of ascertaining Left ventricular contractility and quantifying the correlations in different settings will allow for more accurate and efficient clinical utilization of dp/dtmax in a larger number of clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective cardiac surgical procedures where invasive arterial pressure monitoring and intra-operative transesophageal echocardiography are planned parts of the intra-operative management.
* Age ≥ 18

Exclusion Criteria:

* Age < 18
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective cardiac surgical procedures
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
dp/dt correlations | During the operative period (approximately 5 hours)
  The correlation between dp/dtmax as calculated by the Hypotension Prediction Index (HPI) software and dp/dtmax as calculated by TEE mitral regurgitation jet analysis.

SECONDARY OUTCOMES:
Contractility correlations | During the operative period (approximately 5 hours)
  Determine the correlation between dp/dtmax and standard methods of 2-dimensional and 3-dimensional left ventricular ejection fraction measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Fleming, MD, PhD, Principal Investigator — UC Davis Schoolo of Medicine
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected de-identified patient data
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Completion of enrollment and data analysis
Access Criteria: Contact PI

REFERENCES:
- [Background] Bargiggia GS, Bertucci C, Recusani F, Raisaro A, de Servi S, Valdes-Cruz LM, Sahn DJ, Tronconi L. A new method for estimating left ventricular dP/dt by continuous wave Doppler-echocardiography. Validation studies at cardiac catheterization. Circulation. 1989 Nov;80(5):1287-92. doi: 10.1161/01.cir.80.5.1287. PMID 2805264
- [Background] De Hert SG, Robert D, Cromheecke S, Michard F, Nijs J, Rodrigus IE. Evaluation of left ventricular function in anesthetized patients using femoral artery dP/dt(max). J Cardiothorac Vasc Anesth. 2006 Jun;20(3):325-30. doi: 10.1053/j.jvca.2005.11.006. Epub 2006 Feb 21. PMID 16750731
- [Background] Ostadal P, Vondrakova D, Kruger A, Janotka M, Naar J. Continual measurement of arterial dP/dtmax enables minimally invasive monitoring of left ventricular contractility in patients with acute heart failure. Crit Care. 2019 Nov 21;23(1):364. doi: 10.1186/s13054-019-2654-8. PMID 31752966